CLINICAL TRIAL: NCT05457855
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM) - Montelukast vs Fluticasone
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019P003607-10
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Montelukast: Exposure group
  Interventions: Drug: Montelukast
- Fluticasone: Reference group
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Montelukast — Montelukast claim is used as the exposure group.
  Groups: Montelukast
Drug: Fluticasone — Fluticasone claim is used as the reference group.
  Groups: Fluticasone

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/1u8YFpnMHI5HprhyuY14tIgd1COZcsAWKFlbYCT7aL_A/edit?usp=sharing or Appendix A (https://drive.google.com/file/d/1uC_G8TJ1ujoJbas1p1gFaYFzY7Hw7xMq/view?usp=sharing) for full code and algorithm definitions.

Medicare timeframe: 2008 to 2018 (end of data availability).

Inclusion Criteria:

* 1. Aged >/= 65 years on the index date
* 2. No prior use of Montelukast and Fluticasone anytime prior to cohort entry date
* 3. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date
* 4. At least two claims with asthma diagnosis measured 365 days prior to drug init

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. Prior history of nursing home admission in the 365 days prior to the cohort entry date

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing Montelukast versus Fluticasone. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (cohort entry/index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 51533 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Montelukast | Fluticasone
Started | 12575 | 38958
Completed | 12572 | 12572
Not Completed | 3 | 26386

BASELINE CHARACTERISTICS:
Population: Study cohort after 1:1 propensity score matching
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast | Fluticasone | Total
Number analyzed (Participants) | 12572 | 12572 | 25144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 12572 | 12572 | 25144
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (6.1) | 72.8 (6.1) | 72.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8878 | 8808 | 17686
  Male | 3694 | 3764 | 7458
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10613 | 10650 | 21263
  Black | 831 | 881 | 1712
  Hispanic | 218 | 203 | 421
  Other | 910 | 838 | 1748
Dementia risk factors [Count of Participants; unit: Participants]
  Diabetes | 4098 | 4087 | 8185
  Obesity | 2804 | 2808 | 5612
  Coronary artery disease | 3338 | 3264 | 6602
  Hypertension | 9867 | 9909 | 19776
  Anxiety | 2235 | 2234 | 4469
  Bipolar disorder | 126 | 120 | 246
  Schizophrenia | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Time to Dementia Onset
Description: Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.
Time Frame: Median follow up times: 1) 161 days (exp), 120 days (ref) 2) 504 days (exp), 638 days (ref) 3) 212 days (exp), 130 days (ref) 4) 162 days (exp), 120 days (ref)
Measure: Number (95% Confidence Interval); unit: Incidence rate per 1000 person year
Arm/Group | Montelukast | Fluticasone
Number analyzed (Participants) | 12569 | 12569
Incidence rate per 1000 person year
  Analysis 1 | 9.1 [7.3 to 11.1] | 5.6 [4.0 to 7.7]
  Analysis 2 | 14.5 [12.1 to 17.2] | 14.2 [11.9 to 16.7]
  Analysis 3 | 11.4 [8.7 to 14.9] | 8.6 [5.8 to 12.4]
  Analysis 4 | 3.5 [2.4 to 4.8] | 1.8 [0.97 to 3.1]

ADVERSE EVENTS:
Time Frame: 'As-treated' follow-up approach - Median follow-up days of 161 (for Montelukast) and 120 (for Fluticasone)
Description: Our study did not capture Serious Adverse Events.
Arm/Group | Montelukast | Fluticasone
All-Cause Mortality (participants affected / at risk) | 0/12569 | 0/12569
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/12569 | 0/12569

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT05457855/Prot_SAP_001.pdf